CLINICAL TRIAL: NCT04398862
Title: Measures of Pulmonary Health in Children With Down Syndrome
Brief Title: Pulmonary Health in Children With Down Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-2092; R21HL151261-01 (NIH)
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Down Syndrome; Dysphagia, Oropharyngeal
Keywords: oscillometry; spirometry; outcomes
MeSH Terms: conditions — Down Syndrome; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Down syndrome and aspiration: Outcomes will be compared between two groups although no intervention is submitted, this is an observational study.
- Children with Down syndrome without aspiration: Outcomes will be compared between two groups although no intervention is submitted, this is an observational study.

SUMMARY:
The goal of the study is to learn more about tests that can assess lung health in children with Down syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 18 years, inclusive, at time of consent
* Diagnosis of Down syndrome/trisomy 21 or mosaicism
* Able to walk
* Had a swallow study (video fluoroscopic swallow study or fiberoptic endoscopic evaluation of swallowing) performed within 5 years of consent date

Exclusion Criteria:

* Pregnant or lactating
* Nonambulatory
* Have a tracheostomy or other known severe glottic or subglottic obstruction that would significantly affect the results of testing
* Have a significant acute respiratory illness, defined as treatment with steroids, antibiotics, or an increase in supplemental oxygen
* have a medical illness that would a)increase the risk the participate would incur by participating in the study, b) interfere with the outcomes of the study, or c) interfere with the performance of study participants
* Have a severe behavioral problem that would interfere with the performance of study procedures

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 3-18 years (inclusive) with a diagnosis of Down syndrome who have had a swallow study in the previous 5 years
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-08-21 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Total airway resistance | Baseline
  Airway resistance (R5) measured using forced oscillation technique at 5 Hertz
Airway reactance | Baseline
  Airway reactance (X5) measured using forced oscillation technique at 5 Hertz

SECONDARY OUTCOMES:
Change in total airway resistance after albuterol | Baseline
  Airway resistance (R5) measured using forced oscillation technique at 5 Hertz before and after administration of albuterol
Change in airway reactance after albuterol | Baseline
  Airway reactance (X5) measured using forced oscillation technique at 5 Hertz before and after administration of albuterol
Health-related quality of life, as measured by the Pediatric Quality of Life Inventory | Baseline
  The Pediatric Quality of Life Inventory (PedsQL) assesses four domains of quality of life. Results are converted to a score from 0-100, where low numbers are low quality of life and higher numbers is better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Emily DeBoer, MD, MSCS, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No